CLINICAL TRIAL: NCT04589130
Title: Trial Evaluating Effectiveness of Contrave (Naltrexone HCl / Bupropion HCl) for Weight Maintenance in Adults With BMI ≥ 27 Kg/m2, After 6 Month Intensive Behavior Modification Program: Contrave Obesity Trials (COR) Weight Maintenance Study
Brief Title: Evaluating Contrave for Weight Maintenance in Adults With BMI >= 27 Kg/m2, After 6 Month Behaviour Modification Program.
Acronym: COR-WM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Bausch Health, Canada Inc. (Unknown)
Responsible Party: Principal Investigator, Tony Chetty, Associate Professor Pathology and Molecular Medicine, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR Weight Maintenance Study
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Obesity
Keywords: weight loss maintenance
MeSH Terms: conditions — Obesity | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Intervention Model Description: Parallel - 2 arms during first 6 month phase (treatment and placebo control)
  Crossover - placebo control group crosses over to treatment arm during second 6 months of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking during first 6 month phase (treatment or placebo control).
  All participants receive treatment (Contrave) during second 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contrave 8mg/90mg Extended Release Tablet (Experimental): Group treated with Contrave Extended Release Tablets.
  Interventions: Drug: Contrave 8Mg-90Mg Extended-Release Tablet
- Placebo (Placebo Comparator): Group given placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Contrave 8Mg-90Mg Extended-Release Tablet — Each Contrave Extended Release Tablet contains 8Mg of naltrexone HCl and 90Mg of bupropion HCl and will be administered orally. Total daily dose is 32Mg / 360Mg.
  Participants randomized to the treatment arm will be administered 4 Contrave tablets a day for 1 year (2 tablets taken twice a day).
  Participants randomized to the control arm for the first 6 months will crossover and be administered 4 Contrave tablets a day during the second 6 months (2 tablets taken twice a day). All participants will be in the treatment group (Contrave) during the second 6 month phase of the study.
  Other Names: naltrexone HCl/bupropion HCl
  Arms: Contrave 8mg/90mg Extended Release Tablet
Drug: Placebo — Placebo tablets will be administered orally. Participants randomized to the control arm will be administered 4 placebo tablets a day (2 tablets, taken twice a day) during the first 6 months of the study. These participants will crossover to treatment with Contrave for the second 6 months of the study.
  Other Names: Inactive
  Arms: Placebo

SUMMARY:
Contrave (naltrexone HCl and bupropion HCl) extended-release tablet is an approved drug and indicated to be used with a low calorie diet and increased physical activity for chronic weight management in obese adults (BMI 30 Kg/m2 or greater) or overweight adults (BMI 27 Kg/m2 or greater) with at least one weight related condition such as hypertension or diabetes. Presently we do not have any evidence for the use of Contrave for weight maintenance.

The purpose of this study is to demonstrate that in participants who have ≥ 5% weight loss following the completion of a behaviour modification program with meal replacements, Contrave combined with usual care (dietary and behaviour counselling) will significantly improve maintenance of weight loss and promote further weight loss, compared to placebo with usual care.

DETAILED DESCRIPTION:
Obesity is associated with increased mortality and morbidity and represents a worldwide epidemic that is increasing in prevalence and remains a significant problem in Canada and a burden on our healthcare system. Maintaining long-term weight loss is the "Achilles' heel" of obesity therapy. Since obesity is considered a chronic disease, we need better interventions than continued calorie restriction and increased physical activity.

Sustained weight loss during the first year is a predictive factor for successful weight loss after 4 years. Clinical trials employing an intensive lifestyle intervention demonstrate that a 5-10% weight loss translates into important reductions in metabolic and cardiovascular risk factors. This benefit however, is quite often mitigated by weight regain which could occur in approximately 50% of patients after 1 year. Further behaviour modification/lifestyle intervention and or pharmacotherapy are the main pillars for treating weight regain or achieving weight maintenance. This study will refine our knowledge and understanding about the most appropriate treatment for weight maintenance.

Contrave (naltrexone HCl and bupropion HCl) extended-release tablet is an approved drug and indicated to be used with a low calorie diet and increased physical activity for chronic weight management in obese adults (BMI 30 Kg/m2 or greater) or overweight adults (BMI 27 Kg/m2 or greater) with at least one weight related condition such as hypertension or diabetes. Presently we do not have any evidence for the use of Contrave for weight maintenance.

This is a 1 year, phase 4, prospective, pragmatic, randomized, double-blind, placebo controlled and crossover, observational study that will be conducted in two 6 month phases, across multiple Bariatric Centres of Excellence (BCoE) in Ontario. The first 6 months is the randomized, double blind, placebo controlled phase and participants will be randomly assigned to receive Contrave with usual care (dietary and behaviour counselling) or placebo with usual care. At 6 months and the end of the blinded phase, all participants will be administered Contrave for the remaining 6 month, open-label phase of the study. In other words, participants randomly allocated to receive Contrave will continue on Contrave for the final 6 months, and participants randomly assigned to placebo will crossover to treatment with Contrave for the final 6 months. All subjects will also continue to receive usual care.

The study includes several follow up visits to assess safety and treatment effects, some in person and others by telephone or video conferencing. Body weight, blood pressure, heart rate, waist circumference, lab tests, and subject completed questionnaires will be collected as part of usual care or for the study. Changes in medications and any possible side effects will also be monitored during the study.

To qualify, men and women must successfully complete the BCoE behaviour modification program and demonstrate ≥ 5% weight loss. All participants will be followed for 1 year with multiple visits to assess safety and treatment effects.

This study aims to demonstrate that in participants who have ≥ 5% weight loss following the completion of a behaviour modification program with meal replacements, Contrave combined with usual care will significantly improve maintenance of weight loss and promote further weight loss, compared to placebo with usual care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Body Mass Index (BMI) of ≥ 27 Kg/m2 and the presence of at least one weight related co-morbidity
* Completed 6 month BCoE behaviour modification program with meal replacements and achieved ≥ 5% weight loss since start of program
* Able and willing to provide signed informed consent

Exclusion Criteria:

* Previous surgical treatment for obesity (excluding liposuction if performed more than one year before trial entry)
* History of major depressive disorder or a PHQ-9 (Patient Health Questionnaire-9) score of more than 15 within the last 2 years or history of other severe psychiatric disorders
* Lifetime history of a suicide attempt or history of any suicidal behavior within the past month before entry into the trial
* Pregnancy, planned pregnancy in the next 18 months and or breastfeeding
* Does not agree to use highly effective method of birth control if a woman of child bearing potential, for the duration of the study
* Simultaneous or planned use of other weight loss medication (e.g. Saxenda / Orlistat)
* Uncontrolled hypertension, severe hepatic impairment, end-stage renal disease
* Myocardial infarction or stroke within 6 months prior to consent
* Renal impairment defined as eGFR < 60
* Seizure disorder or a history of seizures or following conditions that may predispose subjects to risk of seizure: history of head trauma, arteriovenous malformation, central nervous system tumor or infection, or a metabolic disorder that in opinion of the investigator may contraindicate treatment with Contrave and increase risk of seizure (e.g. hypoglycemia, hyponatremia)
* Use of other bupropion-containing products (including, but not limited to, Wellbutrin, Wellbutrin SR, Wellbutrin XL, and Zyban), because the incidence of seizure is dose dependent
* A current or prior diagnosis of bulimia or anorexia nervosa, because of a higher incidence of seizures
* Chronic opioid or opiate agonist (eg, methadone) or partial agonists (eg, buprenorphine) use, or acute opiate withdrawal
* Excessive use of alcohol or sedatives, addiction to cocaine or stimulants (street drugs), or withdrawal from sedatives
* Patients undergoing an abrupt discontinuation of alcohol, benzodiazepines or other sedatives and antiepileptic drugs
* Concomitant administration of monoamine oxidase inhibitors (MAOI) (At least 14 days should elapse between discontinuation of a MAOI and initiation of treatment with Contrave.)
* Concomitant administration of the antipsychotic thioridazine, since bupropion may inhibit thioridazine metabolism, thus causing an increase in thioridazine levels and a potential increased risk of thioridazine-related serious ventricular arrythmias and sudden death
* Known hypersensitivity (or known allergic reaction) to the investigational product(s) or any of its ingredients including lactose
* Current participation in another interventional clinical trial
* Not able to complete subject reported, self administered questionnaires or cannot fully understand all instructions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Percentage Change in Body Weight | Week 0 to Week 28
  To determine the weight loss maintenance and any further weight loss effect of Contrave with usual care compared to placebo with usual care, in a post behaviour modification program population.
Percentage of participants who maintained their weight | Week 0 to Week 28
  To determine the weight loss maintenance effect of Contrave with usual care compared to placebo with usual care, in post behaviour modification program population (Participants who had a weight regain less than or equal to 3% of weight from Week 0 - 28 will be regarded as maintainers).
Percentage of participants who lost more than of equal to 5% of body weight | Week 0 to Week 28
  To determine any further weight loss effect of Contrave with usual care compared to placebo with usual care, in a post behaviour modification program population.

SECONDARY OUTCOMES:
Mean Percentage Change in Body Weight from baseline to week 52 | Week 0 to Week 52
  To determine the weight loss maintenance and any further weight loss effect of Contrave compared to placebo, in a post behaviour modification program population.
Percentage of participants who maintained their weight | Week 0 to Week 52
  To determine the weight loss maintenance effect of Contrave compared to placebo, in a post behaviour modification program population (Participants who had a weight regain less than or equal to 3% of weight from Week 0 - 52 will be regarded as maintainers).
Percentage of participants who lost more than or equal to 5% of body weight | Week 0 to Week 52
  To determine any further weight loss effect of Contrave compared to placebo, in a post behaviour modification program population.
Percentage of participants who lost more than or equal to 10% of body weight | Week 0 to Week 28 and Week 52
  To determine any further weight loss effect of Contrave compared to placebo, in a post behaviour modification program population.
Percentage of participants with weight regain (≥ 5% from baseline) | Week 0 to Week 28 and Week 52
  To determine any weight regain in participants taking Contrave compared to placebo, in a post behaviour modification program population.
Percentage of subjects with weight regain (≥ 10% from baseline) | Week 0 to Week 28 and Week 52
  To determine any weight regain in participants taking Contrave compared to placebo, in a post behaviour modification program population.
Mean Percentage Change in Body Weight in participants who crossed over from placebo to Contrave | Week 28 to Week 52
  To determine any weight loss or maintenance effect of Contrave following placebo control phase.
Change in blood pressure (both systolic and diastolic) | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on hypertensive control, in a post behaviour modification program population.
Change in fasting lipid profile | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on total cholesterol, triglycerides, HDL and LDL, in a post behaviour modification program population.
Change in fasting blood glucose | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on diabetes control, in a post behaviour modification program population.
Changes in impulsivity behaviours from baseline as assessed by UPPS-P Impulsive Behaviour Scale (self administered questionnaire) | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on impulsivity behaviours, in a post behaviour modification program population. Urgency, Premeditation (lack of), Perserverance (lack of), Sensation Seeking, Positive Urgency (UPPS-P Impulsive Behaviour Scale)
Changes in quality of life and health economic outcomes. | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on quality of life and health economic outcomes, in a post behaviour modification program population. Assessed by EQ-5D-5L questionnaire.
Percentage of participants who are adherent to pharmacotherapy | Week 0 to Week 28 and Week 52
  To determine the tolerability of Contrave compared to placebo, in a post behaviour modification program setting.
Average number of days participants took investigational product (Contrave or placebo) | Week 0 to Week 28 and Week 52
  To determine the tolerability of Contrave compared to placebo, in a post behaviour modification program setting.
Change in heart rate | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on heart rate, in a post behaviour modification program population.
Change in HbA1c | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on diabetes control, in a post behaviour modification program population.
Changes in eating behaviours from baseline as assessed by Eating Disorder Examination Questionnaire (EDE-Q 6.0) (self administered questionnaire) | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on eating behaviours, in a post behaviour modification program population.
Changes in eating behaviours from baseline as assessed by Yale Food Addiction Scale (YFAS) (self administered questionnaire) | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on eating behaviours, in a post behaviour modification program population.
Changes in food cravings from baseline as assessed by Favourite Food Craving Scale (FFCS) (self administered questionnaire) | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on food cravings, in a post behaviour modification program population.
Changes in depression from baseline as assessed by Patient Health Questionnaire 9 (PHQ-9) (self administered questionnaire) | Week 0 to Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on depression and depressive problems, in a post behaviour modification program population.
Changes in risk of suicidality from baseline as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | Week 0 to Week 12, Week 28 and Week 52
  To determine the effect of Contrave compared to placebo on risk of suicidality, in a post behaviour modification program population.

OTHER OUTCOMES:
Incidences of adverse events (AE) | Week 0 to Week 52
  To determine the safety profile of Contrave in a weight loss maintenance setting in a post behaviour modification population.
Incidences of serious adverse events (SAE) | Week 0 to Week 52
  To determine the safety profile of Contrave in a weight loss maintenance setting in a post behaviour modification population.
Number of participants discontinuing investigational product due to AE/SAEs | Week 0 to Week 52
  To determine the tolerability profile of Contrave in a weight loss maintenance setting in a post behaviour modification program population.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Chetty, MD, Principal Investigator — The Research Institute at St Joseph's Hamilton
Locations (3):
- Canada (3):
  - Guelph General Hospital, Guelph, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No